CLINICAL TRIAL: NCT04981795
Title: realMIND: A Multicenter, Observational Study to Characterize the Safety and Effectiveness of Tafasitamab in Combination With Lenalidomide in US Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma With a Focus on Racial and Ethnic Minority Patients
Brief Title: realMIND: Observational Study on Safety and Effectiveness of Tafasitamab in Combination With Lenalidomide in Patients With Relapsed or Refractory DLBCL
Acronym: realMIND
Status: Recruiting | Type: Observational
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MOR208C414
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — tafasitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Group 1: Racial and ethnic minority patients (at least 50 patients)
  Interventions: Drug: Tafasitamab
- 2: Group 2: Non Hispanic White (NHM) patients (at least 50 patients)
  Interventions: Drug: Tafasitamab

INTERVENTIONS:
Drug: Tafasitamab — Observational Study on safety and effectiveness of tafasitamab in combination with lenalidomide inPatients With Relapsed or Refractory DLBCL.

SUMMARY:
The realMIND study is a multicenter, observational study intended to further characterize the safety and effectiveness data of US patients (with a focus on racial and ethnic minority patients) with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL), treated with tafasitamab in combination with lenalidomide.

DETAILED DESCRIPTION:
This observational study is intended to further characterize the safety and effectiveness of tafasitamab, in combination with lenalidomide, in patients with R/R DLBCL in the US, with a focus on racial and ethnic minorities.

This study also characterizes the overall treatment patterns (e.g., line of treatment, dose modification, combination partners, use as monotherapy) of US patients with R/R DLBCL who have been treated with tafasitamab with a focus on racial and ethnic minorities This multicenter real-world study will help to characterize the use of tafasitamab (e.g., line of treatment, dose modification, combination partners, use as monotherapy) among US patients with R/R DLBCL with a focus on racial and ethnic minorities This is an observational study; as such, no study visits or assessments, laboratory tests or procedures are mandated by the study. Patients will be evaluated and treated according to the physician's usual practice and discretion.

Patient data for this observational study will be collected in one of two ways; either

* by prospective follow-up of patients included at study sites, or
* by retrospective collection of data from patient records, at study sites or from vendor databases.

ELIGIBILITY:
Criteria: Inclusion Criteria:

1. Age ≥18 years at the time of diagnosis of R/R DLBCL
2. Initiated or initiating tafasitamab treatment
3. R/R DLBCL patients who have received at least one (1) prior line of treatment for DLBCL
4. Histologically confirmed DLBCL such as:

   a) DLBCL not otherwise specified (NOS) b) T-cell histiocyte-rich large B-cell lymphoma (THRLBCL) c) Epstein-Barr virus (EBV)-positive DLBCL of the elderly d) Composite lymphoma with a DLBCL component with a subsequent DLBCL relapse, according to Revised European American Lymphoma (REAL)/World Health Organization (WHO) classification e) Patients with evidence of histological transformation to DLBCL from an earlier diagnosis of low-grade lymphoma (i.e., an indolent pathology such as follicular lymphoma [FL], marginal zone lymphoma [MZL], chronic lymphocytic leukemia [CLL]) with a subsequent DLBCL relapse f) High-grade B-cell lymphoma: i) DLBCL with MYC and BCL2 or BCL6 translocation (double-hit) and MYC and BCL2 and BCL6 translocations (triple-hit) ii) High-grade B-cell lymphoma, NOS
5. Signed and dated ICF by the patient or the patient's Legally Acceptable Representative (LAR), for patients with prospective data collection, as applicable. For deceased or otherwise unreachable patients, no informed consent will be obtained for data collection in the study, provided that the competent Independent Ethics Committee (IEC)/Institutional Review Board (IRB) has provided favorable opinion and that any other local regulatory requirements on this matter are met

Exclusion Criteria:

• Initiated or initiating tafasitamab treatment in the context of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Study- 40 sites across the USA
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Patterns - Safety | 2 Years
  Incidence and severity of Treatment-emergent serious AEs (SAEs) and AEs (TEAs)
Treatment Patterns - Effectiveness (a) | 2 Years
  Objective response rate (ORR)
Treatment Patterns - Effectiveness (b) | 2 Years
  Complete response (CR) rate
Treatment Patterns - Effectiveness (c) | 2 Years
  Duration of response (DoR)
Treatment Patterns - Effectiveness (d) | 2 Years
  OS
Treatment Patterns - Effectiveness (e) | 2 Years
  Progression-free survival (PFS)
Treatment Patterns - Effectiveness (f) | 2 Years
  Event-free survival (EFS)

SECONDARY OUTCOMES:
Physician-reported clinical outcome (a) | 2 Years
  Number of treatment lines prior to receiving tafasitamab
Physician-reported clinical outcome (b) | 2 Years
  Distribution of treatment regimens by lines of therapy prior to and subsequent to tafasitamab treatment Duration of tafasitamab treatment (regardless of concomitant treatment with lenalidomide)
Physician-reported clinical outcome (c) | 2 Years
  Duration of combination treatment (i.e., duration of treatment with both tafasitamab and lenalidomide)
Physician-reported clinical outcome (d) | 2 Years
  Modifications of dose and treatment schedule of tafasitamab and/or lenalidomide
Physician-reported clinical outcome (e) | 2 Years
  Incidence of tafasitamab use with combination partners other than lenalidomide
Physician-reported clinical outcome (f) | 2 Years
  Incidence of tafasitamab use as monotherapy (i.e., without any combination partners)

CONTACTS AND LOCATIONS:
Overall Officials: John P Galvin, MD, Study Director — Incyte Corporation
Locations (25):
- United States (25):
  - Alabama Oncology, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - University of California, Irvine Medical Center, Orange, California
  - McFarland Clinic P.C., Ames, Iowa
  - Mission Cancer and Blood, Des Moines, Iowa
  - Tulane Cancer Center, New Orleans, Louisiana
  - American Oncology Partners of Maryland PA, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Westchester Medical Center, Hawthorne, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - VA Medical Center - Durham, Durham, North Carolina
  - Leo Jenkins Cancer Center/ECU School of Medicine, Greenville, North Carolina
  - Mercy Medical Center, Canton, Ohio
  - Ohio Health Marion Area Physicians, Marion, Ohio
  - Tri County Hematology & Oncology Associates, Inc, Massillon, Ohio
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - UW Medicine, Seattle, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Froedtert & Medical College Clinics, Milwaukee, Wisconsin

REFERENCES:
- [Background] Salles G, Duell J, Gonzalez Barca E, Tournilhac O, Jurczak W, Liberati AM, Nagy Z, Obr A, Gaidano G, Andre M, Kalakonda N, Dreyling M, Weirather J, Dirnberger-Hertweck M, Ambarkhane S, Fingerle-Rowson G, Maddocks K. Tafasitamab plus lenalidomide in relapsed or refractory diffuse large B-cell lymphoma (L-MIND): a multicentre, prospective, single-arm, phase 2 study. Lancet Oncol. 2020 Jul;21(7):978-988. doi: 10.1016/S1470-2045(20)30225-4. Epub 2020 Jun 5. PMID 32511983
- [Background] Duell J, Maddocks KJ, Gonzalez-Barca E, Jurczak W, Liberati AM, De Vos S, Nagy Z, Obr A, Gaidano G, Abrisqueta P, Kalakonda N, Andre M, Dreyling M, Menne T, Tournilhac O, Augustin M, Rosenwald A, Dirnberger-Hertweck M, Weirather J, Ambarkhane S, Salles G. Long-term outcomes from the Phase II L-MIND study of tafasitamab (MOR208) plus lenalidomide in patients with relapsed or refractory diffuse large B-cell lymphoma. Haematologica. 2021 Sep 1;106(9):2417-2426. doi: 10.3324/haematol.2020.275958. PMID 34196165
- [Background] Duell J, Abrisqueta P, Andre M, Gaidano G, Gonzales-Barca E, Jurczak W, Kalakonda N, Liberati AM, Maddocks KJ, Menne T, Nagy Z, Tournilhac O, Kuffer C, Bakuli A, Amin A, Gurbanov K, Salles G. Tafasitamab for patients with relapsed or refractory diffuse large B-cell lymphoma: final 5-year efficacy and safety findings in the phase II L-MIND study. Haematologica. 2024 Feb 1;109(2):553-566. doi: 10.3324/haematol.2023.283480. PMID 37646664
- See also: realMIND: Observational Study on safety and effectiveness of tafasitamab in combination with lenalidomide in Patients With Relapsed or Refractory DLBCL (realMIND) — https://www.incyteclinicaltrials.com/study/?id=MOR208C414&SearchTerm=MOR208C414&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=